CLINICAL TRIAL: NCT05360004
Title: The Use of Chinese Herbal Medicine and Vitamin C by Hospital Care Workers in Hong Kong Mobile Cabin Hospital to Prevent COVID-19 Transmission: A Prospective, Randomized Controlled Trial
Brief Title: The Use of Chinese Herbal Medicine and Vitamin C by Hospital Care Workers in HK to Prevent COVID-19
Acronym: CHM-Cov-19-RCT
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hong Kong Baptist University (Other)
Responsible Party: Principal Investigator, ZhaoXiang Bian, Professor, Hong Kong Baptist University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: REC/21-22/0458
Record Dates: First submitted 2022-04-27; First posted 2022-05-04 (Actual); Last update posted 2022-05-04 (Actual); Status verified 2022-05

CONDITIONS: COVID-19
Keywords: Chinese herbal medicine; Prevention; Health Care Worker
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Randomized, open-labelled, controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CHM+Vc (Experimental): Participants in CHM+VC group are required to consume vitamin C 1000mg/day and 1 sachet (9 g) of granules daily (1 hour after meal by dissolving 1 sachet of 9g granules in 150 ml of hot water and drink it orally) .
  Interventions: Drug: Chinese herbal medicine
- Vc (Placebo Comparator): Participants will receive vitamin C 1000mg/day for 14 days
  Interventions: Drug: Chinese herbal medicine

INTERVENTIONS:
Drug: Chinese herbal medicine — CHM is in the form of granules (9 g/sachet), which is comprised of 10 commonly used medicinal herbs: Codonopsis Radix, Astragali Radix, Lonicerae Japonicae Flos, Saposhnikovia Radix, Schizonepetae Herba, Mori Folium, Poria, Atractylodis Rhizoma, Atractylodis Macrocephala Rhizoma, Glycyrrhizae Radix et Rhizoma.

SUMMARY:
This is a prospective randomized controlled trial study to explore whether the combination of Chinese herbal medicine and Vitamin C is effective and safe to prevent COVID-19 transmission among health care workers in Hong Kong Mobile Cabin Hospital governed by the Hong Kong Hospital Authority who have been caring for patients with COVID-19. A total of 652 adults will be enrolled. Eligible subjects who provide written informed consent will be assessed for inclusion/exclusion criteria.

All participants are asymptomatic and test negative for SARS-CoV-2 at the study's commencement. Subjects with major medical illness, renal insufficiency and hypersensitivity to Chinese herbal medicine will be excluded. All participants will receive Vitamin C (VC) supplementation and 28 packets of the herbal medicine free of charge and are advised to consume daily for 14 days. After written informed consent, the subjects will be included and randomly allocated to either CHM+VC group or VC treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Health care workers in Hong Kong Mobile Cabin Hospital;
2. Asymptomatic and test negative for SARS-CoV-2;
3. Aged ≥18;
4. Voluntarily signing a written informed consent form;

Exclusion Criteria:

1. With major medical illness or renal insufficiency;
2. With hypersensitivity to Chinese herbal medicine;
3. Pregnancy or lactation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 652 (Estimated)
Dates: Start 2022-05 (Estimated); Primary Completion 2022-05 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects who become SARS-CoV-2 positive | 4 weeks

SECONDARY OUTCOMES:
Number of days of confirmed SARS-CoV-2 infection | 4 weeks
Duration of COVID-19-related symptoms in confirmed SARS-CoV-2 infection cases | 4 weeks
Safety endpoint | 4 weeks
  Proportion of subjects with treatment-emergent adverse events (TEAEs) and severity of TEAEs (TEAEs are defined as those that are not present at baseline or represent the exacerbation of a pre-existing condition).

IPD SHARING:
Plan to Share IPD: Undecided
All participant data will be de-identified.